CLINICAL TRIAL: NCT02913742
Title: A Prospective Study of the Utility of Neurophysiologic Intraoperative Monitoring by Stereotactic Depth Electrodes During MRI-guided Laser-interstitial Thermal Therapy for Refractory Mesial Temporal Lobe Epilepsy
Brief Title: The Utility of NIOM During LITT for Refractory MTLE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB determined need for an IDE, which was not approved
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00074452
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2016-08

CONDITIONS: Epilepsy, Temporal Lobe
Keywords: Intraoperative Neurophysiological Monitoring
MeSH Terms: conditions — Epilepsy, Temporal Lobe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- monitoring by depth electrode (Experimental): Subjects will be drawn from refractory mesial temporal lobe epilepsy patients determined to be candidates for LITT. During their LITT surgery, in addition to the placement of the stereotactic LITT probe, subjects will receive a second smaller stereotactic electrode for intraoperative monitoring of epileptic discharges before and after surgery. After surgery, at regularly scheduled follow-ups, patients will receive a QOLIE-31-P questionnaire, in addition to standard post-operative care.
  Interventions: Procedure: monitoring by depth electrode

INTERVENTIONS:
Procedure: monitoring by depth electrode — During laser interstitial thermal ablation (LITT) for mesial temporal lobe epilepsy, the study patients will receive invasive neurophysiologic intraoperative monitoring. In addition to the typical placement of LITT stereotactic laser ablation probe via occipital burr hole, the study patients will receive an 8-contact depth recording electrode placed through an adjacent burr hole. The recording electrode will be placed into the parahippocampal gyrus in parallel to the LITT device. The patient will be monitored for epileptic discharges for 10 minutes before and 10 minutes after the ablation process to record the change in discharges during the surgery. The monitoring will not be used to guide surgery. The probe will be removed with the LITT device at the end of the procedure.

SUMMARY:
Mesial temporal lobe epilepsy (MTLE) is the most common cause of medication-resistant epilepsy in adults, and MRI-guided laser interstitial thermal therapy is a new approach to its surgical management; however, while LITT demonstrates fewer complications than traditional surgical techniques, it generates lower rates of seizure freedom. During traditional temporal lobectomy for MTLE, neurophysiologic intraoperative monitoring (NIOM) can be used to better identify epileptogenic tissue and guide resection. Our study proposes to investigate the utility of NIOM during LITT for MTLE. Subjects will be drawn from refractory mesial temporal lobe epilepsy patients determined to be candidates for LITT. During their LITT surgery, in addition to the placement of the stereotactic LITT probe, subjects will receive a second smaller stereotactic electrode for intraoperative monitoring of epileptic discharges before and after surgery. After surgery, at regularly scheduled follow-ups, patients will receive the Quality of Life in Epilepsy questionnaire (QOLIE-31-P), in addition to standard post-operative care. Endpoints will be surgical complications, fractional decrement in epileptiform discharges from pre- to post-ablation recordings, and surgical outcome at 6 months and one year. Analysis of severe complications will be expressed as a simple complication rate, for overall complications, severe complications, and hemorrhagic complications in specific. The relationship between fractional discharge decrement and outcome will be assessed by regression analysis. Risks of the study will stem from the placement of the stereotactic electrode for intraoperative monitoring, which represents a small incremental risk beyond typical LITT for MTLE.

DETAILED DESCRIPTION:
Mesial temporal lobe epilepsy (MTLE) is the most common cause of medication-resistant epilepsy in adults. The standard treatment for refractory MTLE is surgical resection by craniotomy. Stereotactic laser interstitial thermal therapy (LITT) is a new surgical technique being used to treat MTLE. Under MRI-guidance, a laser probe is inserted into the seizure focus and heat is used to destroy the tissue. Compared to temporal lobectomy, LITT results in shorter hospital stays, low complication rates, and possibly less cognitive decline; however, seizure freedom rates are potentially lower.

During temporal lobectomy, neurophysiologic intraoperative monitoring (NIOM) can be used to better identify epileptogenic tissue and guide resection. This tool has been unavailable during LITT procedures. Recently, the investigators demonstrated in two cases that NIOM with a depth electrode is technically feasible during LITT and can identify epileptiform activity intra-operatively.

This is a prospective trial of NIOM during LITT for mesial temporal lobe epilepsy. The investigators will assess the safety of performing NIOM during LITT and whether data from NIOM (frequency and characteristics of epileptiform discharges recorded before and after ablation) are associated with seizure outcomes. If there is an association, NIOM could be used for prognostication and could potentially even be used to guide surgery.

Hypotheses:

1. NIOM performed by MRI-guided stereotactic depth electrode placed in the parahippocampal gyrus adjacent to the LITT catheter is safe, as compared to institutional LITT controls without NIOM and published LITT complication rates.
2. Greater magnitude fractional decrements in discharge frequency from pre-ablation to post-ablation recordings will be significantly associated with better seizure outcomes, as measured by International League Against Epilepsy (ILAE) surgical outcome scores.

Objectives:

The primary project goals are to assess if NIOM by parahippocampal depth electrode is safe during LITT of MTLE and to assess if the fractional decrement of interictal discharges (ID) on NIOM can be significantly correlated with outcome. The study will be powered to address these questions a priori. Post hoc analyses consisting of a multivariate analysis of other patient demographic data, NIOM findings, operative parameters, quality of life scores, and neuropsychiatric outcomes will also be assessed.

ELIGIBILITY:
Inclusion criteria are as follows

1. Age ≥ 18
2. The patient must suffer from drug resistant mesial temporal lobe epilepsy as determined by a consensus of providers at weekly epilepsy surgery conferences held by the Duke Epilepsy Center
3. The patient must be a candidate for LITT for MTLE as determined by a consensus of providers at weekly epilepsy surgery conferences held by the Duke Epilepsy Center

Exclusion criteria are as follows

1. Age ≤ 18
2. Lack of consensus on localization of MTLE
3. Multifocal epilepsy
4. History of prior epilepsy surgery
5. Lack of consensus on candidacy for LITT
6. Pregnancy
7. Patient without capacity to provide legal consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
fractional decrement in interictal epileptiform discharges (ID) from pre- to post-ablation | 30 day post-operative course
  Analysis of NIOM ID recordings will focus on fractional decrement of discharge counts from pre- to post-operative recordings. Fractional decrement was chosen, as opposed to absolute discharge counts, which are expected to vary widely among patients. Fractional discharge decrement will be assessed for its association with surgical outcome.
Surgical complications associated with intraoperative monitoring electrodes and recording | Perioperative through 30 days post-operation
  Analysis of safety will occur in an ongoing fashion, and at completion of the trial. Major complications will be reviewed immediately per institutional review board (IRB) approved protocols, and will trigger a project safety evaluation. Moderate and minor complications will be recorded, with results reviewed quarterly, to assess project safety. Final safety results will be compared to registry data of institutional MTLE LITT procedures and to published LITT results for MTLE.

SECONDARY OUTCOMES:
Epilepsy surgery outcome | Perioperative through 30 days post-operation
  Outcome will be measured by the ILAE surgical outcome 6-point scale. Fractional ID decrement will be analyzed for their association with surgical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Luedke, MD, Principal Investigator — Duke University Hospital
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Luedke MW, Pietak MR, Serafini S, Haglund MM, Sinha SR. Intraoperative ECoG During MRI-Guided Laser-Interstitial Thermal Therapy for Intractable Epilepsy. J Clin Neurophysiol. 2016 Aug;33(4):e28-30. doi: 10.1097/WNP.0000000000000299. PMID 27261642